CLINICAL TRIAL: NCT00605436
Title: Restorative Yoga for Therapy of the Metabolic Syndrome: A Pilot Trial
Brief Title: Yoga for the Treatment of Metabolic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Cliff Lede Foundation (Unknown)
Responsible Party: Alka M. Kanaya, MD
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H9377-29543-02; CHR#H9377-29543-02
Record Dates: First submitted 2008-01-16; First posted 2008-01-31 (Estimated); Last update posted 2008-01-31 (Estimated); Status verified 2008-01

CONDITIONS: Metabolic Syndrome
Keywords: overweight; sedentary; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Restorative yoga therapy group: one orientation workshop for 3 hours, then twice-weekly group yoga therapy classes for first 5 weeks followed by once-weekly group yoga classes for another 5 weeks. The group will also be asked to practice their yoga postures at home for 30 minutes three times per week.
  Interventions: Behavioral: Restorative yoga therapy
- B (No Intervention): The control group is a wait-list control group with no active intervention.

INTERVENTIONS:
Behavioral: Restorative yoga therapy — 3-hour workshop at study initiation. Then twice-weekly group yoga classes for 5 weeks, then once-weekly group yoga classes for 5 weeks. Home yoga practice for 90 minutes/week throughout the 10 week trial.
  Arms: A

SUMMARY:
We tested the following hypotheses:

1. That a standardized yoga therapy will improve insulin sensitivity (primary outcome), and other features of the metabolic syndrome such as hypertension and dyslipidemia (secondary outcomes), we will perform a 2-hour oral glucose tolerance test, fasting blood tests, and a physical examination before and after randomization of subjects to a 10-week yoga therapy intervention or wait-list control group.
2. That a yoga therapy is feasible in overweight and underactive individuals with the metabolic syndrome, that adherence to a yoga intervention is acceptable, and that yoga therapy is associated with improved quality of life, we will assess the adherence to twice-weekly yoga group sessions (for weeks1-5) and weekly yoga group sessions (for weeks 6-10), frequency of home yoga therapy practice, and self-reported quality of life before and after the intervention in both treatment groups.
3. To elucidate a potential mechanism for the effect of yoga on changes in insulin resistance by evaluating markers of inflammation from adipose tissue (adipocytokines). We hypothesize that these biochemical parameters will show modest improvement with yoga therapy and that changes in these parameters will be associated with improvements in insulin sensitivity.

DETAILED DESCRIPTION:
Study Interventions: There will be a 12-week intervention period.

1. Yoga Therapy Group: Those randomized to yoga therapy will receive twice-weekly group yoga sessions at the Osher Center for the entire intervention period. The yoga postures and breathing techniques will be taught by a qualified and certified yoga instructor using a standardized protocol that was determined by a Yoga Expert Panel. Each group yoga session will take approximately 90 minutes. Participants will also be required to practice yoga at home at least 3 times per week, and be given yoga materials (mat, blocks, straps), an instruction manual, and a video for their use at home. They will be asked to keep a calendar log of the dates/times that they practiced yoga at home. This group will also receive a 20-30 minute session with a counselor to discuss Standard Health Education at the beginning of the 12-week intervention. This session will be similar to the control group intervention.
2. Standard Health Education Group: Participants assigned to the standard health education group will receive an individual 20-30 minute session with a trained research associate within a week of their baseline visit. In this session, participants will be informed of the importance of a healthy lifestyle, given written information of the Food Guide Pyramid12 and told to follow the equivalent of the National Cholesterol Education Program Step I diet13. They will be counseled to reduce weight and increase physical activity. This is similar to the intervention given to the "Standard Lifestyle Group" in the Diabetes Prevention Program4.

ELIGIBILITY:
Inclusion Criteria:

1. to be between the ages of 30 and 65 years,
2. fulfill at least three criteria for the metabolic syndrome per the NCEP guidelines:

   * waist circumference (>88 cm for women; >102 cm for men),
   * HDL-cholesterol (<50 mg/dl for women; <40 mg/dl for men),
   * triglycerides >=150 mg/dL
   * fasting glucose >=100 mg/dL, and/or
   * high blood pressure (>=130/>=85 or use of antihypertensive medication), and
3. report an underactive or sedentary lifestyle defined as accumulating less than 30 minutes of moderate intensity endurance exercise 5 days per week.

Exclusion Criteria:

1. Pregnancy or lactation
2. Coronary heart disease (defined as a myocardial infarction or cardiac intervention with percutaneous transluminal catheterization or coronary artery bypass graft surgery) event or hospitalization in the past 6 months
3. Chronic illnesses: cancer, kidney disease, cirrhosis, rheumatogic diseases, or chronic infections
4. Current use of these medications: oral diabetes medications, insulin, steroid hormones, oral contraceptives, hormone replacement therapy, niacin, fibrates.
5. Regular participation (>1/week) yoga for past 3 months or concurrent use of yoga
6. Current major psychiatric illness, cognitive impairment, or substance abuse
7. Plans to move out of the study region within 6 months
8. Life-expectancy of < 6 months
9. Concurrent enrollment in any other studies, experimental therapies, or blinded treatments

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose level | 10 weeks

SECONDARY OUTCOMES:
Feasability of yoga postures | 10 weeks
Adherence to protocol | 10 weeks
Blood pressure | 10 weeks
Insulin sensitivity | 10 weeks
Weight | 10 weeks
Waist circumference | 10 weeks
Heart rate variability | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alka M. Kanaya, MD, Principal Investigator — University of California, San Francisco; Deborah Grady, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States